CLINICAL TRIAL: NCT03643107
Title: Phase II Study of Irofulven in AR-targeted and Docetaxel-Pretreated Metastatic Castration-Resistant Prostate Cancer Patients, Who Have a Drug Response Predictor (DRP®) Indicating a High Likelihood of Response to Irofulven.
Brief Title: Irofulven in AR-targeted and Docetaxel-Pretreated mCRPC Patients With Drug Response Predictor (DRP®)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allarity Therapeutics (Industry)
Collaborators: Smerud Medical Research International AS (Other); Lantern Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMR-3165; 2017-003549-72 (EudraCT Number)
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer Patients
Keywords: Drug Response Prediction (DRP)
MeSH Terms: interventions — irofulven; Prednisolone

STUDY DESIGN:
Intervention Model Description: Irofulven will be administered as an intravenous dose of 0.45 mg/kg, over a 30-minute infusion period by venous access at day 1 and 8 of a three week cycle.
  Irofulven will be administered in combination with a daily dose of 10 mg orally administered prednisolone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irofulven + Prednisolone 10mg (Experimental): Irofulven will be administered as an intravenous dose of 0.45 mg/kg, over a 30-minute infusion period by venous access at day 1 and 8 of a three week cycle.
  Irofulven will be administered in combination with a daily dose of 10 mg orally administered prednisolone.
  Interventions: Drug: Irofulven; Combination Product: Prednisolone 10 mg

INTERVENTIONS:
Drug: Irofulven — Irofulven will be administered as an intravenous dose of 0.45 mg/kg, over a 30-minute infusion period by venous access at day 1 and 8 of a three week cycle.
  Irofulven will be administered in combination with a daily dose of 10 mg orally administered prednisolone.
Combination Product: Prednisolone 10 mg — Irofulven will be administered as an intravenous dose of 0.45 mg/kg, over a 30-minute infusion period by venous access at day 1 and 8 of a three week cycle.
  Irofulven will be administered in combination with a daily dose of 10 mg orally administered prednisolone.

SUMMARY:
The study seek to evaluate the anti-tumor effect after treatment of Irofulven in combination with prednisolone in patients who progressed on androgen receptor(AR)-targeted therapy and Docetaxel-Pretreated Metastatic Castration-Resistant Prostate Cancer Patients. A drug response predictor (DRP®) biomarker in prostate cancer patients will identify patients likely to respond to and benefit from treatment with Irofulven.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically confirmed adenocarcinoma or poorly differentiated carcinoma of the prostate (carcinomas with pure small-cell histology or pure high grade neuroendocrine histology are excluded; neuroendocrine differentiation is allowed)
* Surgically or medically castrated, with serum testosterone levels of ≤ 50 ng/dL. For patients currently being treated with luteinizing hormone-releasing hormone (LHRH) agonists, i.e., patients who have not undergone an orchiectomy, therapy must be continued throughout the study
* Have evidence of disease progression after prior therapy for mCRPC:
* Disease progression after treatment with at least 1 but no more than 2 prior next-generation AR-targeted therapies (abiraterone acetate, enzalutamide, or investigational AR-targeted agent) for metastatic prostate cancer (treatment with the older anti-androgen therapies such as bicalutamide, flutamide, and nilutamide are not counted toward this limit), AND
* Disease progression after treatment with docetaxel for metastatic prostate cancer. Prior Docetaxel therapy administered for hormone-sensitive disease is permitted and is not counted toward this limit
* Disease progression after initiation of most recent therapy is based on any of the following criteria:
* Rise in PSA: a minimum of 2 consecutive rising levels, with an interval of ≥ 1 week between each determination. The most recent screening measurement must have been ≥ 1 ng/mL
* Transaxial imaging: new or progressive soft tissue masses on CT or MRI scans as defined by RECIST 1.1
* Radionuclide bone scan: at least 2 new metastatic lesions
* Signed informed consent obtained prior to initiation of any study-specific procedures or treatment.
* Age ≥ 18 years
* Life expectancy ≥ 3 months
* Performance status 0 - 1
* Have participated in the Irofulven screening protocol in which the Drug Response Predictor (DRP) outcome is measured as being in the upper limit of response (defined as being in the top 20%). Scaling can be modified depending on the clinical outcome.
* Adequate organ functions
* Hematological: absolute neutrophil count (ANC) >1.5 x 10E9/L, platelet count >100 x 10E9/L, hemoglobin ≥ 6.2 mmol/L
* Hepatic: Bilirubin within normal range, aspartate transaminase (AST) and alanine transaminase (ALT) ≥ 2.5 upper normal limit (UNL), albumin > 25 g/L
* Renal: creatinine clearance ≥ 30 mL/min (calculated according to the Cockcroft and Gault method)
* Recovered to grade 0 or 1 from any toxic effects of prior chemotherapy, radiotherapy

Exclusion Criteria:

* Prior external beam radiation therapy to >25% of the bone marrow
* Contraindication to the use of prednisolone (e.g. uncontrolled diabetes mellitus)
* Prior treatment with Irofulven.
* Ongoing treatment with a corticosteroid at a prednisolone-equivalent dose > 10 mg/day
* More than 1 prior treatment with either isotopes Sm or Sr, or radioisotope treatment or treatment with bisphosphonate agents or antibody treatment i.e., denosumab within 2 months prior to initiation of treatment with investigational Medicinal Product (IMP). Pre-existing treatment with bisphosphonate agents or denosumab is to be continued during the study
* Initiation of treatment with bisphosphonate agents or antibody treatment i.e., denosumab, within 4 weeks of study start. Pre-existing treatment with bisphosphonate agents or denosumab is to be continued during the study
* Treatment with coumarin derivatives and/or phenytoin most be discontinued and coagulation parameters most be within the normal range before treatment with Irofulven
* History of significant gastric or small bowel resection, malabsorption syndrome, or other lack of integrity of the upper gastrointestinal tract that may prevent compliance with oral drug administration
* Presence of any serious concomitant systemic disorders and/or psychiatric condition incompatible with the study (at the investigators discretion)
* History of retinopathy
* Presence of any active infection (at the investigators discretion).
* Central Nervous System Disease (CNS) disease including epilepsy or altered mental status precluding understanding of the informed consent process and/or completion of the necessary study procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Anti-tumor effect of Irofulven with prednisolone | one year
  Objective response rate defined as complete response, partial response or stable disease > 9 weeks according to RECIST 1.1 for patients with measurable disease and defined as stable disease > 9 weeks according to Prostate Cancer Working Group 3 (PCWG3) for bone metastases

SECONDARY OUTCOMES:
Duration of response (DOR) | one year
  Time from documentation of tumor response to disease progression
Radiologic progression free survival (rPFS) | one year
  rPFS defined as ≥ two new lesions on an 8-week bone scan plus two additional lesions on a confirmatory scan, ≥ two new confirmed lesions on any scan ≥ 9 weeks after enrolment, and/or progression in nodes or viscera on cross-sectional imaging, or death.
Overall survival | one year
  Time from enrolment until death from any cause.
Prostate Specific Antigen (PSA) response | one year
  ≥ 50% decline in PSA compared to baseline in all patients according to PCWG3
PSA response | one year
  ≥ 90% decline in PSA compared to baseline in all patients according to PCWG3
Time to PSA progression | one year
  PSA progression defined in accordance with PCWG3.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Dept. Of Oncology, Copenhagen, Denmark